CLINICAL TRIAL: NCT04859660
Title: Pre-operative Tamsulosin After Minimally Invasive Hysterectomy and Time to Spontaneous Void: A Randomized Controlled Trial
Brief Title: Pre-operative Tamsulosin and Time to Spontaneous Void After Hysterectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2102483026
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-06

CONDITIONS: Urinary Retention Postoperative
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamsulosin- intervention group (Experimental)
  Interventions: Drug: Tamsulosin
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — Participants will be given Tamsulosin or placebo in the pre-op bay prior to surgery. Post-operatively, time to void and time to discharge from the post-anesthesia care unit will be recorded.
  Arms: Tamsulosin- intervention group
Drug: Placebo — Participants will be given Tamsulosin or placebo in the pre-op bay prior to surgery. Post-operatively, time to void and time to discharge from the post-anesthesia care unit will be recorded.
  Arms: Placebo group

SUMMARY:
The aim of this study is to determine if a one time dose of tamsulosin given pre-operatively decreases the time to void and the time to discharge after minimally invasive hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-80 undergoing outpatient minimally invasive hysterectomy

Exclusion Criteria:

* Inability to provide informed consent
* Bladder malignancy
* Intra-operative bladder or ureteral injury; anticipated prolonged bladder catheterization
* Plan for sling or anterior repair

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Banner University Medical Center- Phoenix, Phoenix, Arizona
  - Banner University Medical Center- Tucson, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gabra M, Hall C, McCann L, Shah J, Jones I, Masjedi A, Runke S, Hsu CH, Aguirre A. Tamsulosin and Time to Spontaneous Void After Hysterectomy: A Randomized Controlled Trial. Obstet Gynecol. 2024 Dec 1;144(6):810-816. doi: 10.1097/AOG.0000000000005724. Epub 2024 Sep 12. PMID 39265173

RESULTS

PARTICIPANT FLOW:
Groups:
- Tamsulosin- Intervention Group: Tamsulosin arm: Participants will receive a single dose of 0.4mg oral Tamsulosin capsule in the pre-op bay 1-2 hours before surgery.
- Placebo Group: Placebo arm: Participants will receive a single dose of oral placebo capsule in the pre-op bay 1-2 hours before surgery.
Period: Overall Study
Arm/Group | Tamsulosin- Intervention Group | Placebo Group
Started | 81 | 80
Completed | 77 | 73
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Tamsulosin- Intervention Group: Tamsulosin arm: Participants will be given Tamsulosin in the pre-op bay
- Placebo Group: Placebo arm: Participants will be given Placebo the pre-op bay.
- Total: Total of all reporting groups
Arm/Group | Tamsulosin- Intervention Group | Placebo Group | Total
Number analyzed (Participants) | 77 | 73 | 150
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [34 to 46] | 42 [35 to 45] | 41 [34 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 73 | 150
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 15 | 34
  Not Hispanic or Latino | 46 | 47 | 93
  Unknown or Not Reported | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 62 | 54 | 116
  More than one race | 3 | 7 | 10
  Unknown or Not Reported | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 77 | 73 | 150
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 30 [26 to 38] | 31 [26 to 37] | 30 [26 to 38]
Current smoker [Count of Participants; unit: Participants] | 12 | 8 | 20
Parity [Mean (Inter-Quartile Range); unit: Living births] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Charston Comorbidity index [Count of Participants; unit: Participants]
  Score 0 (no health conditions) | 62 | 58 | 120
  Score 1 | 11 | 11 | 22
  Score 2 | 3 | 4 | 7
  Score 3 | 0 | 0 | 0
  Score 4 (several health conditions) | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Spontaneous Void
Description: Each participant underwent a void trial post-operatively by backfilling their bladder with 200cc normal saline at the conclusion of the case and removing the foley. Patients needed to void at least 100cc to be considered to have "passed" their void trial.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Tamsulosin- Intervention Group | Placebo Group
Number analyzed (Participants) | 77 | 73
hours | 1.63 [0.94 to 2.44] | 1.42 [0.84 to 2.33]

2. Secondary Outcome: Time to Discharge From the Post-anesthesia Care Unit
Description: The time from the patient leaving the OR to the time they were discharged home from the Post-anesthesia care unit was recorded to determine the Time to discharge.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Tamsulosin- Intervention Group | Placebo Group
Number analyzed (Participants) | 77 | 73
hours | 2.4 [1.7 to 3.5] | 2.6 [1.9 to 3.5]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Participation in this study involves minimal risk
Arm/Group | Tamsulosin- Intervention Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/80
Serious Adverse Events (participants affected / at risk) | 2/81 | 1/80
Other Adverse Events (participants affected / at risk) | 4/81 | 3/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamsulosin- Intervention Group (N=81) | Placebo Group (N=80)
Hospital admission (Cardiac disorders) | 0 (0) | 1 (1) — Exacerbation of heart failure
Vaginal cuff dehiscence (Reproductive system and breast disorders) | 2 (2) | 0 (0) — Vaginal cuff dehiscence
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamsulosin- Intervention Group (N=81) | Placebo Group (N=80)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Pelvic abscess (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Emergency room visit for gastritis
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1) — Emergency room visit for kidney stones
vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Emergency room visit for vaginal bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT04859660/Prot_SAP_001.pdf